CLINICAL TRIAL: NCT05096715
Title: Phase IB Study of Atezolizumab and Bevacizumab With SBRT for Unresectable Hepatocellular Carcinoma
Brief Title: Atezolizumab+Bevacizumab+SBRT in Unresectable HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-286
Record Dates: First submitted 2021-08-30; First posted 2021-10-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — atezolizumab; Bevacizumab; Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Stereotactic beam radiation therapy (SBRT) +Atezolizumab + Bevacizumab (Experimental): Study will begin with a safety lead of 6 participants to determine the maximum tolerated dose (MTD) of Stereotactic beam radiation therapy (SBRT) with atezolizumab and bevacizumab followed by study expansion to 14 more participants after maximum tolerated dose (MTD) is established.
  Safety Lead-In: 6 cycles/18 weeks (study cycle is 3 weeks/21 days)
  * Cycle 1: Atezolizumab + Bevacizumab (1x) with Stereotactic beam radiation therapy (SBRT) every 1-3 days
  * Cycles 2-6: Atezolizumab + Bevacizumab (1x) every 3 weeks
  Expanded Study:
  * Cycle 1: Atezolizumab + Bevacizumab (1x) with Stereotactic beam radiation therapy (SBRT) every 1-3 days
  * Cycles 2-End:Atezolizumab + Bevacizumab (1x) every cycle
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Radiation: Stereotactic body radiation therapy (SBRT)

INTERVENTIONS:
Drug: Atezolizumab — Intravenous Infusion
  Other Names: Tecentriq
Drug: Bevacizumab — Intravenous Infusion
  Other Names: Mvasi; Zirabrev
Radiation: Stereotactic body radiation therapy (SBRT) — External Beam Radiation
  Other Names: Radiation Therapy

SUMMARY:
This research study is evaluating the safety and tolerability of the drugs atezolizumab and bevacizumab with stereotactic body radiation therapy (SBRT) for treating unresectable hepatocellular carcinoma.

This study involves the following interventions:

* Atezolizumab
* Bevacizumab
* Stereotactic body radiation therapy (SBRT)

DETAILED DESCRIPTION:
This is a single-arm phase 1B study designed to evaluate the combination of Atezolizumab and Bevacizumab with stereotactic body radiation therapy (SBRT for treating and limiting the recurrence of unresectable hepatocellular carcinoma.

The U.S. Food and Drug Administration (FDA) has approved atezolizumab and bevacizumab for unresectable hepatocellular carcinoma. The FDA has not approved the combination of radiation therapy, atezolizumab, and bevacizumab.

Atezolizumab is believed to work by increasing the immune system's response to cancer cells. Bevacizumab is believed to work by inhibiting cancer cells from growing by targeting a specific protein in the cancer cells. Radiation therapy is a standard of care treatment for unresectable hepatocellular carcinoma. Radiation therapy has also been shown to increase the effects of drugs like atezolizumab and bevacizumab.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will be in this research study for as long as the study drugs are safe and beneficial to them. Participants will then be followed for up to 5 years.

It is expected that about 20-32 people will take part in this research study.

Genentech, a biotechnology company, is supporting this research study by providing funding for the study, including the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have diagnosis of hepatocellular carcinoma (HCC) that is deemed unsuitable for surgical resection, transplant, or radiofrequency ablation (RFA). Participants may have up to 5 lesions with a total maximal tumor dimension of < 20 cm, and no one lesion > 15 cm. Diagnosis may be confirmed by at least 1 criteria listed below:

  * Histologically or cytologically proven diagnosis of HCC within 180 days prior to study registration.
  * At least 1 solid liver lesion or vascular tumor thrombus (involving portal vein, IVC, and/or hepatic vein) > 1 cm with arterial enhancement and delayed washout on multiphasic CT or MRI. Radiologic imaging evaluation must occur within 28 days prior to study registration.
  * Enhancing vascular thrombosis demonstrating arterial enhancement and delayed washout of multiphasic MRI. Radiologic imaging evaluation must occur within 30 days prior to study registration.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Small volume extrahepatic disease permitted, defined as <2.0 cm in sum of maximal diameters (e.g. presence of one 1.8 cm metastatic lymph node, or two 0.8 cm lung lesions are allowed). Bony lesions are included in the <2.0 cm of extrahepatic disease. Note that benign periportal lymphadenopathy is not unusual in the presence of hepatitis and is permitted, even if the sum of enlarged nodes is > 2.0 cm. Radiologic imaging of chest, abdomen, and pelvis via CT or MRI is required within 28 days prior to study registration. CT with contrast is required unless contrast is contraindicated.
* Participants may have received transarterial chemoembolization (TACE) or drug eluting beads (DEB). A 2 week (14 day) washout period is required prior to initiating study treatment.
* Age ≥18 years at the time of signing informed consent document.
* ECOG performance status 0-1.
* Child-Pugh A liver function within 7 days of study registration.
* Barcelona Clinic Liver Cancer (BCLC) stages Intermediate (B) or Advanced (C) within 7 days of study registration.
* No evidence of significant portal hypertension.
* Participants must have adequate organ and marrow function as defined the following laboratory results, obtained within 7 days prior to study registration:

  * absolute neutrophil count ≥1,500/mcL
  * absolute lymphocyte count ≥500/mcL
  * platelets ≥75,000/mcL without transfusion
  * hemoglobin ≥9 g/dL, transfusion allowed to meet this criterion
  * total bilirubin ≤ 3 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤5 × institutional ULN
  * alkaline phosphatase(ALP) <2 × institutional ULN
  * creatinine ≤ 1.5 × institutional ULN OR
  * estimated creatinine clearance ≥50 mL/min/1.73 m2 (according to the Cockcroft-Gault formula)
  * serum albumin ≥2.8 g/dL
  * INR or aPTT ≤2 × institutional ULN for participants not receiving therapeutic anticoagulation
  * Urine dipstick for proteinuria <2+; participants discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1g of protein in 24 hours.
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade ≤ 1 prior to study entry, with the exception of alopecia.
* No known HIV infection.
* Documented virology status of hepatitis B virus (HBV), as confirmed by screening HBV serology test within 28 days prior to study registration.

  * For participants with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * For participants with active HBV, HBV DNA <500 IU/mL obtained within 28 days prior to initiation of study treatment, and Anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study.
* Documented virology status of hepatitis C virus (HCV), as confirmed by screening HCV serology test within 28 days prior to study registration.
* Women of childbearing potential (WOCBP) must agree to use appropriate method(s) of contraception to avoid pregnancy during the treatment period and for at least 5 months after the last dose of Atezolizumab or 6 months after the last dose of Bevacizumab. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 14 days prior to study registration.
* Women must not be breastfeeding.
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year during the treatment period and for 6 months after the last dose of Bevacizumab. Men must refrain from donating sperm during this same period.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior systemic therapy
* Prior radiation to the region of the liver that would result in excessive doses to normal tissues due to overlap of RT fields is not allowed. Radiotherapy within 28 days and abdominal/pelvic radiotherapy within 60 days prior to initiation of study treatment are not allowed. Exception for palliative radiotherapy to bone lesions within 7 days prior to initiation of study treatment.
* Prior selective internal radiotherapy (SIRT) or hepatic arterial Yttrium therapy, at any time.
* Direct tumor extension into the stomach, duodenum, small bowel, or large bowel.
* Extrahepatic metastases or malignant nodes (that enhance with typical features of HCC) > 2 cm, in sum of maximal diameters (e.g. presence of one 2.4 cm metastatic lymph node or two 1.2 cm lung lesions).
* Known fibrolamellar HCC, sarcomatoid HCC, or biphenotypic HCC.
* History of leptomingeal disease.
* GI bleed within 6 months prior to study registration.
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses (<30 mm from the carina) of large volume. Participants with vascular invasion of the portal or hepatic veins may be enrolled.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment is not allowed. Abdominal surgery, abdominal interventions, or significant abdominal traumatic injury within 60 days prior to initiation of study treatment is not allowed. Participants who have not recovered from side effects of any such procedure are ineligible. Anticipation of need for a major surgical procedure during the study should reconsider enrollment.
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g. <% risk of recurrence or 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, superficial bladder cancer, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g. to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior allogenic stem call or solid organ transplantation.
* Clinically significant bleeding or clotting risk requiring treatment.
* History of hemoptysis (≥2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. Prophylactic anticoagulation for the patency of venous access is allowed provided the activity of the agents results in INR <1.5 x ULN and aPTT is within normal limits within 14 days prior to study registration. Prophylactic use of low molecular-weight heparin (i.e. enoxaparin 40 mg/day) is allowed.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to the first dose of Bevacizumab.
* History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment.
* History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement of routine parenteral hydration, parenteral nutrition, or tube feeding within 6 months prior to initiation of study treatment. Participants with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at the time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for the symptom resolution.
* History of intra-abdominal inflammatory process within 6 months prior to initiation of study treatment, including but not limited to peptic ulcer disease, diverticulitis, or colitis.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during Atezolizumab treatment or within 5 months after the last dose of Atezolizumab. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist.) are live attenuated vaccines, and are not allowed.
* History of severe anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the Atezolizumab or Bevacizumab formulation.
* Patients with untreated or incompletely treated varices with bleeding or high risk for bleeding. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to study registration. Patients who have undergone an EGD within 6 months prior to initiation of study treatment do not need to repeat the procedure.
* Moderate or severe ascites.
* Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure.
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
* History of hepatic encephalopathy.
* Active co-infection of HBV and HCV. Participants with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV.
* Known history of HIV infection.
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan. Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

  * Measurable disease, per RECIST v1.1, must be present outside the CNS.
  * Participant has no history of intracranial hemorrhage or spinal cord hemorrhage.
  * Metastases are limited to the cerebellum or the supratentorial region (i.e. no metastases to the midbrain, pons, medulla, or spinal cord).
  * No evidence of interim progression between completion of CNS-directed therapy and initiation of study treatment.
  * Participant has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, neurosurgical resection within 28 days prior to initiation of study treatment.
* Current or recent (within 10 days of first dose of study treatment) use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
* Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID) with the exception of daily Aspirin 81 mg. Occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed.
* Uncontrolled tumor-related pain. Participants requiring pain medication must be on a stable regimen at study entry.

  * Symptomatic lesions (e.g. bone metastases or metastases causing nerve impingement amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.)
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g. epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Participants with indwelling catheters (e.g. PleurX®) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected serum calcium > ULN)
* Treatment with investigational therapy within 28 days prior to initiation of study treatment.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the initiation of study treatment.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g. 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g. fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) ≥150 mmHg and/or diastolic blood pressure >100 mmHg), based on an average of ≥ 3 BP readings on ≥ 2 sessions. Anti-hypertensive therapy to achieve these parameters is allowable.
* Prior history of hypertensive crisis or hypertensive encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity Rate | 18 weeks
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Progression free survival (PFS) | 5 years
  Assessed per HCC mRECIST, imRECIST, and RECIST v1.1
Overall Survival (OS) | 5 years
  Estimated using the Kaplan-Meier method
In-field response rate | 5 years
  Assessed per RECIST v1.1, imRECIST, and HCC mRECIST
Change in Child-Pugh Score | 2.5 years
  Analyzed as repeated measures using mixed models to characterize the trend over time. Child-Pugh scores range from 5 to 15, with higher scores indicating worse outcomes.
Out of field response rate | 2.5 years
  Assessed per RECIST v1.1, imRECIST and HCC mRECIST among patients with low volume metastatic disease

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Y Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation